CLINICAL TRIAL: NCT01252602
Title: Prospective Study of Maternal Prenatal Depression as a Risk Factor for Failure to Breastfeed
Brief Title: Prenatal Depression and Failure to Breastfeed
Status: Withdrawn | Type: Observational
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Principal Investigator, Pamela McCool, OBGYN, Oklahoma State University Center for Health Sciences
Other Study IDs: 2010-024
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Breastfeeding After Discharge From Hospital Following Childbirth, Yes/no; Depression Scale Score
Keywords: breastfeeding, EPDS, prenatal depression
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prenatally depressed: Women who tested positive for prenatal depression with a score of > 12 on the Edinburgh Postnatal Depression Scale
- Not Prenatally Depressed: Women who tested not depressed on the prenatal depression scale with a score < 13

SUMMARY:
The purpose of this prospective cohort study is to search for a relationship between maternal depression in the third trimester, as indicated by a score of > 12 on the EPDS, and a choice not to breastfeed at all, defined as no breastfeeding after dismissal from the hospital. The investigators hypothesize that women who screen positive for prenatal depression will be significantly less likely to breastfeed their babies after discharge from the hospital following childbirth.

DETAILED DESCRIPTION:
Introduction

Postpartum depression (PPD) is a form of major depressive disorder (MDD) and affects about 15% of mothers following birth (1). This condition is a serious medical matter, not only because of the suffering it causes the women, but because it can negatively affect the infant emotionally, socially, and even cognitively, sometimes far beyond the time of the depression (2). Many physicians now routinely screen for PPD at the traditional 4-6 week postpartum visit, and such screening has been the policy at OSU clinics for the past decade. However, Kim et al (2008) recently reported that testing pregnant women at 24-28 weeks gestation for depression resulted in a risk status that was identical with risk status after delivery for 90% of patients studied (3). The author concluded that prenatal screening for possible later PPD seemed clinically useful.

Various studies have investigated a possible relationship between PPD and failure to breastfeed, with mixed results. Misri et al (1997) reported that 83% of their subjects with PPD experienced onset after discontinuing breastfeeding (4). Henderson et al (2003) reported that a study of 1,745 Australian women revealed that subjects with PPD were more likely to stop breastfeeding than non-depressed ones (5). In addition, they found that the women tended to wean after onset of PPD (5). However, McKee et al (2004) found no association between PPD and beginning or duration of breastfeeding (6). Further, Hatton et al (2005) found that although women with more depressive symptoms were less likely to breastfeed at 6 weeks postpartum than their counterparts without symptoms, this difference could not be found at 12 weeks postpartum (7).

Here at OSU, Dr. Sarah McCoy published two studies on breastfeeding and PPD in 2006 and 2008, both of which were retrospective reviews of records (8, 9). The first one was a more selective and smaller sample than the second, because at the time the data were collected, PPD screening had not quite become universal. In that first study of 209 subjects, a significant relationship was found between breastfeeding and scores above 12 on the Edinburgh Postnatal Depression Scale (EPDS), which indicated PPD (8). However, the second similarly-designed study of 588 subjects, which was a more representative sample of the clinic population, failed to confirm those results (9).

To date, little if any studies have been published that deal directly with the topic of prenatal depression and its relationship to whether a woman chooses to breastfeed after giving birth. However, McCarter-Spaulding and Horowitz (2007) recently recommended prenatal screening for PPD in anticipation of potential roadblocks to breastfeeding (10). If it could be shown that women with prenatal depressive symptoms are less likely to choose breastfeeding, perhaps early intervention could increase the number of infants that are breastfed, which is an important public-health goal (11).

Purpose The purpose of this prospective cohort study is to search for a relationship between maternal depression in the third trimester, as indicated by a score of > 12 on the EPDS, and a choice not to breastfeed at all, defined as no breastfeeding after dismissal from the hospital.

Methods The investigators plan to collect data from women that are receiving prenatal care at the OSU Houston Parke clinic. Upon obtaining informed consent at a prenatal appointment between 34 weeks + 0 days gestation and 37 weeks + 6 days, (should consent be deemed necessary), the investigators will ask the subjects to fill out the same EPDS screen that OSU obstetrics patients already typically fill out at the four-week postpartum appointment. Filling out that scale at a prenatal appointment is the only activity that the test subjects will be asked to do that is not already a standard part of their obstetrics' treatment. In addition, the investigators will note these women's EPDS score at the four-week postpartum visit and whether or not they choose to breastfeed, as well as the other information listed under "Data Collection", most of which are already routinely recorded in the chart.

Early Termination Criteria Patient will also be terminated if they do not follow up at their postpartum visit.

Drugs and Dosages No drugs are used in this project. Devices The only device used in this study is the EPDS. Surgical Procedures This study does not include any surgical procedures. Data Collection

Information recorded for the study will include:

1. Gestational age at prenatal EPDS screen
2. Prenatal EPDS score
3. Use of any antidepressants at the time of the prenatal screening
4. Use of any antidepressants after the prenatal screening
5. Age of patient
6. Whether infant was stillborn yes/no
7. Whether infant had birth defects yes/no
8. Whether infant had illness that prevented breastfeeding
9. Whether infant breastfed at all after leaving the hospital
10. Whether infant was still breastfeeding at the four-week postnatal appointment

Confidentiality Data will be de-identified after the four-week postpartum visit by conversion to numbers. It will be recorded on an Excel spreadsheet.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant female in third trimester obtaining prenatal care through OSU Houston Parke obstetrics clinic 2. All questions of both EPDS assessments completed, one at 34 + 0 days-37 + 6 days weeks gestation and one at the standard four-week postnatal examination 3. Breastfeeding status noted on chart at four-week postpartum examination, yes/no, with yes defined as any activity, exclusive or partial, after dismissal from the hospital

-

Exclusion Criteria:

1. Use of anti-depressive medication after initial prenatal EPDS administration 2. Mothers of stillborn infants, infants with an illness that prevented breastfeeding, or of infants with birth defects 3. Incomplete EPDS questionnaire, either prenatal or postnatal

-

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women receiving prenatal care at the OSU Houston Parke obstetrics clinic in Tulsa, Oklahoma, who are in their third trimester between 34 and 38 weeks gestation
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
EPDS score | late third trimester - four weeks postpartum
  Numerical value on maternal depression screening test

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J McCool, DO, Principal Investigator — Oklahoma State University Center for Health Sciences

REFERENCES:
- [Result] Hatton DC, Harrison-Hohner J, Coste S, Dorato V, Curet LB, McCarron DA. Symptoms of postpartum depression and breastfeeding. J Hum Lact. 2005 Nov;21(4):444-9; quiz 450-4. doi: 10.1177/0890334405280947. PMID 16280561
- [Result] Kim JJ, Gordon TE, La Porte LM, Adams M, Kuendig JM, Silver RK. The utility of maternal depression screening in the third trimester. Am J Obstet Gynecol. 2008 Nov;199(5):509.e1-5. doi: 10.1016/j.ajog.2008.04.018. Epub 2008 Jun 4. PMID 18533122
- [Result] Henderson JJ, Evans SF, Straton JA, Priest SR, Hagan R. Impact of postnatal depression on breastfeeding duration. Birth. 2003 Sep;30(3):175-80. doi: 10.1046/j.1523-536x.2003.00242.x. PMID 12911800
- [Result] McCoy SJ, Beal JM, Shipman SB, Payton ME, Watson GH. Risk factors for postpartum depression: a retrospective investigation at 4-weeks postnatal and a review of the literature. J Am Osteopath Assoc. 2006 Apr;106(4):193-8. PMID 16627773
- [Result] McCoy SJ, Beal JM, Saunders B, Hill EN, Payton ME, Watson GH. Risk factors for postpartum depression: a retrospective investigation. J Reprod Med. 2008 Mar;53(3):166-70. PMID 18441719
- [Result] McCarter-Spaulding D, Horowitz JA. How does postpartum depression affect breastfeeding? MCN Am J Matern Child Nurs. 2007 Jan-Feb;32(1):10-7. doi: 10.1097/00005721-200701000-00004. PMID 17308452